CLINICAL TRIAL: NCT04741633
Title: Multi Dimensional Precise Exploration of Immunoconsolidation Therapy for Locally Advanced Non-small Cell Lung Cancer After Chemo-radiotherapy
Brief Title: Multi Dimensional Precise Exploration of Immunoconsolidation Therapy for Locally Advanced NSCLC After Chemo-radiotherapy
Acronym: NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Dr., Fudan University
Other Study IDs: CID-001
Record Dates: First submitted 2021-01-02; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: NSCLC; Chemoradiotherapy; ctDNA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to carry out a prospective observational study in patients with locally advanced NSCLC receiving radical concurrent chemoradiotherapy and follow-up immune consolidation therapy. By detecting ctDNA and TILs of the patients, we explored the value of blood dynamic monitoring of ctDNA in patients with prognosis stratification and treatment effect, and explored the patients before and after concurrent chemoradiotherapy and immune consolidation therapy The characteristics of DNA, RNA, T cells and other biomarkers were correlated with the efficacy and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Non small cell lung cancer patients confirmed by pathology;
2. They were 18-80 years old;
3. The tumor could not be resected or could not tolerate surgery;
4. Planed to receive chemoradiotherapy and subsequent immunoconsolidation therapy;
5. Clinical stage III (AJCC, 8th Edition, 2017);
6. After systematic detection of non-small cell lung cancer core indicators including EGFR, ALK, ros1, KRAS, ntrk, TMB, etc;
7. Patient informed consent.

Exclusion Criteria:

1. After radiotherapy and chemotherapy, the disease progressed and immune maintenance therapy could not be carried out
2. It can not cooperate with the completion of baseline mutation screening and subsequent sample detection
3. Factors judged by other researchers not suitable for further study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced NSCLC receiving radical concurrent chemoradiotherapy and subsequent immunoconsolidation therapy
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between ctDNA dynamic detection and 1-year PFS rate after chemoradiotherapy | Six months after consolidation treatment
  The ctDNA dynamic detection will contain NGS test including mutations(both somatic and germline), copy number variations, gene fusions along with genetic interpretation for each and every mutation identified in each test(both blood and tissue) during the whole therapeutic process

SECONDARY OUTCOMES:
PFS | Six months after consolidation treatment
OS | Six months after consolidation treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China